CLINICAL TRIAL: NCT06985303
Title: Phase 1 Study Evaluating the Safety and Preliminary Efficacy of a Novel Cell-Based and Small Molecule Combination Therapy for White Matter Injury in Patients With Periventricular Leukomalacia
Brief Title: Cell-Based Therapy for White Matter Repair in Periventricular Leukomalacia
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Based on a review of new preclinical findings, the sponsor has decided to conduct additional foundational research before initiating this clinical study. The study is withdrawn pending further investigation.
Sponsor: MGAM LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGAM-001
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Periventricular Leukomalacia; White Matter Disease; Hypoxic-Ischemic Encephalopathy; Demyelinating Diseases; Neonatal Encephalopathy
Keywords: Periventricular Leukomalacia; Myelin Repair; White Matter Injury; Demyelination; Neonatal Brain Injury; Neuroregeneration; CNS Regeneration; Brain Repair; Neonatal Hypoxia
MeSH Terms: conditions — Leukomalacia, Periventricular; Leukoencephalopathies; Hypoxia-Ischemia, Brain; Demyelinating Diseases; Asphyxia Neonatorum

STUDY DESIGN:
Intervention Model Description: This is a single-group assignment study where all participants receive the investigational therapy. The therapy is a multi-component treatment combining a proprietary cell-based product with several molecular and enzymatic agents. This model allows for an initial assessment of the safety, tolerability, and biological activity of this combination approach for promoting white matter repair in PVL.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental: Investigational Combination Therapy (Experimental): Participants will receive an investigational combination therapy. This therapy consists of a proprietary cell-based component administered with a cocktail of molecular and enzymatic agents. These agents are designed to support cell health, promote myelin repair, and reduce inhibitory factors in the damaged brain tissue. The overall goal of the intervention is to promote white matter regeneration in patients with periventricular leukomalacia by targeting key barriers that prevent natural repair.
  Interventions: Combination Product: Investigational Combination Product

INTERVENTIONS:
Combination Product: Investigational Combination Product — This investigational therapy combines a proprietary, human-derived cell-based component with a unique blend of small molecules and an enzyme. The components are designed to work synergistically to address the complex pathology of white matter injury. The therapy aims to provide a source for cellular regeneration, support the survival of existing cells, enhance the potential for myelin repair, and modify the inhibitory environment of glial scar tissue. This multi-pronged biological intervention is designed to promote neural regeneration and functional recovery in patients with PVL.

SUMMARY:
The goal of this study is to explore a new treatment that may help repair brain damage in individuals with periventricular leukomalacia (PVL), a condition that affects white matter in the brain. Researchers are testing whether a combination of a novel cell therapy and specific molecular agents can support brain repair.

The main questions the study aims to answer are:

Can the treatment help regrow white matter and improve myelin repair? Does the treatment reduce scarring in the brain? Is the treatment safe and well-tolerated?

The study uses several components, including:

A specific type of neural progenitor cell to form the basis of the therapy. A small molecule compound to support cell function and survival. An agent designed to promote the repair of the myelin sheath. An enzyme intended to break down scar tissue in the brain. Researchers will study how these components work together to protect and repair the brain by influencing key pathways involved in damage and recovery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of periventricular leukomalacia (PVL) confirmed by MRI
* Clinically stable at time of intervention
* Parental or legal guardian consent if participant is a minor

Exclusion Criteria:

* Severe congenital brain malformations unrelated to PVL
* Active CNS infection or systemic inflammatory disease
* History of severe intraventricular hemorrhage (Grade III/IV)
* Known allergy or history of a significant hypersensitivity reaction to the investigational product or any of its components.
* Participation in another interventional study within the past 30 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in White Matter Integrity | At baseline and 12 weeks post-intervention
  Measured using fractional anisotropy (FA) values derived from diffusion tensor imaging (DTI) MRI to assess structural white matter characteristics in brain regions affected by periventricular leukomalacia (PVL).

SECONDARY OUTCOMES:
Change in Functional Motor Score | Baseline, 6 weeks, and 12 weeks post-intervention
  Measured using the Gross Motor Function Measure-88 (GMFM-88). The scale ranges from 0 to 100; higher scores indicate better motor function.
Change in Glial Scar Density | 12 weeks post-intervention
  Quantified using established biomarkers for astrogliosis, such as glial fibrillary acidic protein (GFAP), from cerebrospinal fluid or via advanced imaging. This outcome is intended to measure the biological activity of the therapy's scar-reducing component.

IPD SHARING:
Plan to Share IPD: No